CLINICAL TRIAL: NCT02492204
Title: The Role of IL33/ST2 Axis in ARDS Patients
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IL33/ST2
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2018-01

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days

GROUPS / COHORTS (2):
- Survivors
- Non survivors

SUMMARY:
The main objective is the study of the role of IL33/ST2 axis in the pathogenesis of ARDS, it´s value as prognosis marker and as therapeutic target.

ELIGIBILITY:
Inclusion Criteria:

* ARDS
* Risk pathologies to develop ARDS (sepsis, pancreatitis, pneumonia, massive transfussion, politraumatics)

Exclusion Criteria:

* Age under 18
* Pregnancy
* Undergoing a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ARDS criteria according to Berlin definition or risk pathologies
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Actual); Study Completion 2019-12

PRIMARY OUTCOMES:
Prognostic value of the IL-33/ST2 axis in patients with ARDS. | 60 days

SECONDARY OUTCOMES:
Value of IL33/ST2 axis to predict development of ARDS in risk patients | 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitary Vall d´Hebron, Barcelona, Spain